CLINICAL TRIAL: NCT06351488
Title: Detection of Circulating Kidney DNA in Kidney Transplant Patients Facing an Episode of Graft Rejection
Acronym: DART-RREGREF
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CGenetix (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP231661
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant; Rejection
Keywords: Graft rejection; renal circulating DNA; performance of the diagnostic test
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — two additional tubes of blood of 10 mL and 6 mL respectively as well as a urine sample of 22 mL will be collected to mainly measure the quantity of plasma DNA of renal origin circulating in the blood during an episode of graft rejection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In France, 3,500 kidney transplants are carried out per year; and 40,000 people succeed in 2019 with a kidney transplant. Despite regular medical monitoring, nearly 30% of transplant patients will develop rejection. Currently, only solid biopsy of the graft makes it possible to establish the diagnosis of graft rejection, and to characterize its cellular origin based on the Banff classification.

Several studies have shown the possibility of identifying the tissue origin of DNA circulating in the blood, in healthy subjects, on the basis of the epigenetic properties of circulating DNA. In addition, in kidney transplant subjects, an increase in the quantity of circulating DNA originating from the graft in the blood and urine has been shown as well as an increase in urinary chemokine levels during renal dysfunction (notably dismiss). Thus, the company CGenetix in partnership with INSERM units 1155 and 1151 is developing a method to identify and characterize kidney transplant rejection early, through the detection of epigenetic biomarkers on circulating DNA targeting different fractions of the kidney (glomerular, tubular, peritubular capillary and vascular). The main objective is to study the diagnostic performance of the quantity of DNA of renal origin in kidney transplant patients in the blood and in the urine (expressed in copies/ml) for the diagnosis of type Rejection mediated by kidneys. antibody (ABMR) established by kidney graft biopsy (gold standard) and according to the Banff 2022 classification.

DETAILED DESCRIPTION:
Kidney transplantation remains the standard treatment for patients with end-stage renal disease. It provides the patient with a better quality of life1 and a better chance of survival, for a reduced cost of care compared to dialysis. While more than 3,000 kidney transplants are carried out each year in France, more than 20,000 candidates are registered on the transplant waiting list, revealing a severe shortage of grafts. Limiting the degradation of the kidney graft would make it possible to avoid the return of patients to dialysis and limit the shortage of grafts.

At the diagnostic level, routine monitoring of graft functionality after kidney transplantation is based on the use of non-specific markers, such as serum creatinine (allowing the estimation of glomerular filtration rate or GFR) and proteinuria. Definitive diagnosis of renal allograft dysfunction still requires invasive allograft biopsy, which remains the gold standard for evaluating graft status. The anatomopathological diagnosis of renal graft dysfunction is based on the Banff classification, and makes it possible to examine the immune infiltrate and cellular lesions of the graft in order to make a diagnosis on: 1-the presence of graft rejection or other attacks and 2- the anatomical compartment affected by the pathology: tubular, vascular, interstitial or glomerular.

The start-up CGenetix offers an original approach to predict and characterize renal graft rejection/dysfunction based on the quantification of epigenetic signatures present on donor-cell-free DNA. In 2018, Moss et al. are developing a deconvolution model capable of identifying the tissue origin of circulating DNA by taking advantage of its epigenetic properties. The study confirmed that the free DNA circulating in healthy subjects comes mainly from blood cells and endothelial cells, but not from kidney cells.

In this protocol, 319 kidney transplant patients will be recruited from the Renal Transplantation departments of Pitié-Salpêtrière and Necker. Patients will be recruited into the study at the time of their hospitalization for renal biopsy for cause/indication (inclusion visit). Urine and blood samples will be taken within 24 hours before the kidney biopsy is performed.

The quantities of circulating DNA of renal origin (total kidney biomarkers (x2), specific tubules (x2), specific glomeruli (x2), specific peritubular capillaries (x2) and specific arteriolar capillaries (x2)) will be determined by digital PCR and expressed in copy/ml in blood and urine samples.

The main evaluation criterion of the research is the area under the ROC curve of the ABMR type rejection prediction models according to renal biopsy and with as covariates of interest the quantities of circulating DNA of renal origin (kidney biomarkers total (x2), specific tubules (x2), specific glomeruli (x2), specific peritubular capillaries (x2) and specific arteriolar capillaries (x2)) determined by digital PCR and expressed in copy/ml in blood and urine The final objective of this study protocol consists of i) prospectively validating the performance of the diagnostic test proposed by CGenetix and its partners INSERM 1155 and 1151 and urinary chemokines to non-invasively diagnose acute renal graft rejection and ii ) study its ability to diagnose the different types of renal transplant rejection (ABMR, TCMR, Mixed, Without rejection) The research hypotheses are: i) an AUC ≥ 0.80 / Sensitivity and specificity ≥ 80% for each biomarker taken individually; ii) an AUC ≥ 0.85 / Sensitivity and specificity ≥ 85% for the multimodal prediction model.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Patient living with at least one functioning kidney graft
* Summoned to perform a kidney biopsy for cause/indication at the Pitié Salpêtrière Hospital or at the Necker Hospital
* Having been informed of the study and not opposing the study
* Benefiting from a social security system (excluding AME)

Exclusion Criteria:

* Under legal protection measure (curatorship or guardianship, under judicial protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant patients eligible for a solid biopsy
Sampling Method: Non-Probability Sample
Enrollment: 319 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
The area under the ROC curve of ABMR rejection prediction models according to kidney biopsy and with renal circulating DNA quantities as variables of interest | At the time of the biopsy for suspicion of graft rejection
  The probability of ABMR rejection, established by kidney graft biopsy and according to the Banff 2022 classification, will be predicted with logistic regression models which will integrate the number of copies/ml of the 10 genes measured by PCR in blood or urine. and tested individually.

SECONDARY OUTCOMES:
The area under the ROC curve of TCMR rejection prediction models according to kidney biopsy and with renal circulating DNA quantities as variables of interest | At the time of the biopsy for suspicion of graft rejection
  The probability of TCMR rejection, established by kidney graft biopsy and according to the Banff 2022 classification, will be predicted with logistic regression models which will integrate the number of copies/ml of the 10 genes measured by PCR in blood or urine. and tested individually.
The area under the ROC curve of mixed rejection prediction models according to kidney biopsy and with renal circulating DNA quantities as variables of interest | At the time of the biopsy for suspicion of graft rejection
  The probability of mixed rejection, established by kidney graft biopsy and according to the Banff 2022 classification, will be predicted with logistic regression models which will integrate the number of copies/ml of the 10 genes measured by PCR in blood or urine. and tested individually.
The area under the ROC curve of glomerulitis-type rejection prediction models (≥g1) according to kidney biopsy and with renal circulating DNA quantities as variables of interest | At the time of the biopsy for suspicion of graft rejection
  The probability of glomerulitis-type rejection, established by kidney graft biopsy and according to the Banff 2022 classification, will be predicted with logistic regression models which will integrate the number of copies/ml of the 10 genes measured by PCR in blood or urine. and tested individually.
The area under the ROC curve of tubulitis-type rejection prediction models (≥t1) according to kidney biopsy and with renal circulating DNA quantities as variables of interest | At the time of the biopsy for suspicion of graft rejection
  The probability of tubularitis-type rejection, established by kidney graft biopsy and according to the Banff 2022 classification, will be predicted with logistic regression models which will integrate the number of copies/ml of the 10 genes measured by PC
The area under the ROC curve of vascularitis-type rejection prediction models (≥v1) according to kidney biopsy and with renal circulating DNA quantities as variables of interest | At the time of the biopsy for suspicion of graft rejection
  The probability of vascularitis-type rejection, established by kidney graft biopsy and according to the Banff 2022 classification, will be predicted with logistic regression models which will integrate the number of copies/ml of the 10 genes measured by PCR in blood or urine. and tested individually.
The area under the ROC curve of capillaritis-type rejection prediction models (≥ptc1) according to kidney biopsy and with renal circulating DNA quantities as variables of interest | At the time of the biopsy for suspicion of graft rejection
  The probability of capillaritis-type rejection, established by kidney graft biopsy and according to the Banff 2022 classification, will be predicted with logistic regression models which will integrate the number of copies/ml of the 10 genes measured by PCR in blood or urine. and tested individually.
Areas under the ROC curve of rejection prediction models according to renal biopsy and with as covariates of interest the quantities of urinary chemokines (CXCL9 and CXCL10) determined by ELISA and expressed in pg/mL in urine | At the time of the biopsy for suspicion of graft rejection
  The main endpoint of the research is the area under the ROC curve of the ABMR, TCMR, mixed rejection prediction models according to renal biopsy and with the quantities of urinary chemokines (CXCL9 and CXCL10) as covariates of interest. ) determined by ELISA and expressed in pg/mL in urine

CONTACTS AND LOCATIONS:
Overall Officials: Pierre GALICHON, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Assistance Publique - Hôpitaux de Paris, Hôpital Necker, Paris
  - Assistance Publique - Hôpitaux de Paris, Pitié-Salpêtrière hospital, Paris
  - Assistance Publique - Hôpitaux de Paris, Hôpital Tenon, Paris